CLINICAL TRIAL: NCT05467462
Title: The Efficacy of Four Different Treatment Regimes of Uterotonic Agents for Prevention of Postpartum Hemorrhage at Vaginal Delivery: A Multicentric Randomized Controlled Trial
Brief Title: Efficacy of Four Different Treatment Regimes on Postpartum Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 04.07.2022-E.69157
Record Dates: First submitted 2022-07-18; First posted 2022-07-20 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Postpartum Hemorrhage
Keywords: postpartum hemorrhage; oxytocin; carbetocin; tranexamic acid
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin; Oxytocin; Tranexamic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Carbetocin (Experimental): 100-mg carbetocin was intravenously administered immediately after birth of the baby
  Interventions: Drug: I.V carbetocin administration
- Oxytocin Group (Experimental): The oxytocin infusion consisting of 20 IU dissolved in 500 mL of normal 0.9 % sodium chloride solution and infused at a rate of 125 mL/h was administered immediately after clamping the umbilical cord
  Interventions: Drug: I.V Oxytocin administration
- Carbetocin and Tranexamic acid Group (Experimental): 100-mg carbetocin was intravenously administered immediately after birth of the baby and tranexamic acid infusion consisting of 1gr dissolved in 100 mL of normal 0.9 % sodium chloride solution was administered immediately after clamping the umbilical cord
  Interventions: Drug: I.V carbetocin and tranexamic acid administration
- Oxytocin and Tranexamic acid Group (Experimental): The oxytocin infusion consisting of 20 IU dissolved in 500 mL of normal 0.9 % sodium chloride solution and infused at a rate of 125 mL/h was administered and tranexamic acid infusion consisting of 1gr dissolved in 100 mL of normal 0.9 % sodium chloride solution was administered immediately after clamping the umbilical cord
  Interventions: Drug: I.V Oxytocin and tranexamic acid administration

INTERVENTIONS:
Drug: I.V carbetocin administration — Group I: carbetocin was intravenously administered immediately after birth of the baby.
  Other Names: carbetocin
  Arms: Carbetocin
Drug: I.V Oxytocin administration — Group II: Oxytocin the oxytocin infusion consisting of 20 IU dissolved in 500 mL of normal 0.9 % sodium chloride solution and infused at a rate of 125 mL/h was administered immediately after clamping the umbilical cord.
  Other Names: Oxytocin
  Arms: Oxytocin Group
Drug: I.V carbetocin and tranexamic acid administration — Group III: carbetocin and tranexamic acid 100-mg carbetocin was intravenously administered immediately after birth of the baby and tranexamic acid infusion consisting of 1gr dissolved in 100 mL of normal 0.9 % sodium chloride solution was administered immediately after clamping the umbilical cord.
  Other Names: carbetocin and tranexamic acid
  Arms: Carbetocin and Tranexamic acid Group
Drug: I.V Oxytocin and tranexamic acid administration — Group IV: oxytocin and tranexamic acid the oxytocin infusion consisting of 20 IU dissolved in 500 mL of normal 0.9 % sodium chloride solution and infused at a rate of 125 mL/h was administered and tranexamic acid infusion consisting of 1gr dissolved in 100 mL of normal 0.9 % sodium chloride solution was administered immediately after clamping the umbilical cord
  Other Names: Oxytocin and tranexamic acid
  Arms: Oxytocin and Tranexamic acid Group

SUMMARY:
Postpartum hemorrhage is the most important cause of maternal morbidity and mortality worldwide and accounts for approximately 25% of deaths worldwide. Drugs such as oxytocin, carbetocin and tranexamic acid are used for bleeding control after normal vaginal delivery. The most widely used agent for the prevention of postpartum hemorrhage worldwide is oxytocin. The primary aim of this study is to reduce the mean blood loss after vaginal delivery. In this study, investigators aimed to compare the efficacy of carbetocin alone in the 1st group, oxytocin alone in the 2nd group, carbetocin and tranexamic acid in the 3rd group, and oxytocin and tranexamic acid in the 4th group in preventing postpartum blood loss originating from the uterus.

DETAILED DESCRIPTION:
This prospective, randomized controlled study was conducted at the Department of Obstetrics and Gynecology of Bezmialem University Hospital and Van Regional Training and Research Hospital between August 2022 and February 2023. The study protocol was approved by the Ethical Committee of the Medical Faculty of Bezmialem University. Written informed consent was obtained from all patients. Investigators included a total of 272 women between 18 and 40 years of age who came to hospital for vaginal delivery at term single pregnancy. This trial was designed and reported according to the Consolidated Standards of Reporting Trials (CONSORT) guidelines.

The patients included in this study were randomly divided into four groups by random allocation using a computer-generated random number. Group I: carbetocin (Pabal®; Ferring Pharma, Istanbul, Turkey) (n = 68 )(was intravenously administered immediately after birth of the baby). Group II: Oxytocin(Synpitan forte®; Deva Pharma, Istanbul, Turkey) (n =68)(the oxytocin infusion consisting of 20 IU dissolved in 500 mL of normal 0.9 % sodium chloride solution and infused at a rate of 125 mL/h was administered immediately after clamping the umbilical cord) Group III: carbetocin and tranexamic acid (Transamin; TEVA Pharma, Istanbul, Turkey)2 (n =68) (100-mg carbetocin was intravenously administered immediately after birth of the baby and tranexamic acid infusion consisting of 1gr dissolved in 100 mL of normal 0.9 % sodium chloride solution was administered immediately after clamping the umbilical cord) . Group IV: oxytocin and tranexamic acid (n=68) (the oxytocin infusion consisting of 20 IU dissolved in 500 mL of normal 0.9 % sodium chloride solution and infused at a rate of 125 mL/h was administered and tranexamic acid infusion consisting of 1gr dissolved in 100 mL of normal 0.9 % sodium chloride solution was administered immediately after clamping the umbilical cord).The collected data were age, prepregnancy body mass index (BMI), gravida, parity, gestational age at birth, Apgar scores at 1 and 5 min, birth weight, neonatal intensive care unit (NICU) admission, the prepartum hemoglobin and hematocrit concentrations, the change in the hemoglobin and hematocrit concentrations (difference between prepartum and postpartum levels), duration of delivery stages, intrapartum blood loss and estimated blood loss after 2 hours of vaginal delivery.

In this study, the investigators aimed to compare the efficacy of oxytocin, carbetocin and tranexamic acid in preventing uterine blood loss during vaginal delivery.

ELIGIBILITY:
Inclusion Criteria

* Single pregnancy greater than 37 weeks
* Pregnant women between the ages of 18-40
* Volunteer

Exclusion Criteria:

* Pregnancy less than 37 weeks
* Patients under stress who cannot give informed consent
* Patients allergic to carbetocin, oxytocin or tranexamic acid
* Clinical diagnosis of a serious cardiovascular disease
* Clinical diagnosis of severe liver disease
* Clinical diagnosis of kidney disease
* Clinical diagnosis of epilepsy
* Internal feature with risk for embolism or bleeding
* Refusing to volunteer

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 300 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Hemogram status | Postpartum 24th hour
  Postpartum hemogram status

SECONDARY OUTCOMES:
Blood Transfusion | Postpartum 24th hour
  Number of patients needing Blood Transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Gurkan Kıran, MD, Study Chair — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Grotegut CA, Paglia MJ, Johnson LN, Thames B, James AH. Oxytocin exposure during labor among women with postpartum hemorrhage secondary to uterine atony. Am J Obstet Gynecol. 2011 Jan;204(1):56.e1-6. doi: 10.1016/j.ajog.2010.08.023. Epub 2010 Nov 3. PMID 21047614
- [Result] Chard T, Boyd NR, Forsling ML, McNeilly AS, Landon J. The development of a radioimmunoassay for oxytocin: the extraction of oxytocin from plasma, and its measurement during parturition in human and goat blood. J Endocrinol. 1970 Oct;48(2):223-34. doi: 10.1677/joe.0.0480223. No abstract available. PMID 5471863
- [Result] Hunter DJ, Schulz P, Wassenaar W. Effect of carbetocin, a long-acting oxytocin analog on the postpartum uterus. Clin Pharmacol Ther. 1992 Jul;52(1):60-7. doi: 10.1038/clpt.1992.103. PMID 1623693